CLINICAL TRIAL: NCT07043517
Title: TEMPOROMANDIBULAR JOINT DYSFUNCTION IN CHILDREN WITH CEREBRAL PALSY: ASSOCIATIONS WITH GMFCS LEVELS, SUBTYPES, AND BRUXISM
Brief Title: TMJ Dysfunction and Motor Severity in Children With CP
Status: Completed | Type: Observational
Sponsor: Istanbul Arel University (Other)
Collaborators: Kayseri University (Other)
Responsible Party: Principal Investigator, Ozge Baykan Copuroglu, Asst. Prof., Istanbul Arel University
Other Study IDs: TMDCPPrevalance; YOK-Tez-ID:896940 (Other: Mugla Sıtkı Kocman University)
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy; Temporomandibular Disorder (TMD)
Keywords: cerebral palsy; temporomandibular joint; GMFCS
MeSH Terms: conditions — Cerebral Palsy; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cerebral palsy: GMFCS Level 1-4
  Interventions: Other: RDC/TMD

INTERVENTIONS:
Other: RDC/TMD — TMJ functions were assessed using the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD).

SUMMARY:
This study aims to examine the function of the temporomandibular joint (TMJ)-the jaw joint-in children with cerebral palsy (CP). Children with CP often experience difficulties in jaw movement, pain, or involuntary grinding of teeth (bruxism), which can affect their ability to eat, speak, or smile comfortably.

The research will investigate how the severity of motor impairment, as classified by the Gross Motor Function Classification System (GMFCS), and different CP subtypes are related to jaw function problems. The study also explores the relationship between bruxism and TMJ pain and dysfunction.

By performing clinical evaluations of mouth opening, jaw movements, muscle tenderness, and pain levels, this study hopes to identify early signs of TMJ problems. The goal is to provide better recommendations for early screening, therapy, and rehabilitation for children with CP, especially those with more severe motor impairments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cerebral palsy (CP) by a pediatric neurologist, based on standard clinical criteria.
* Aged between 6 and 18 years.
* Classified as GMFCS Levels I to IV.
* Able to comply with clinical assessment procedures.
* Written informed consent obtained from parent(s) or legal guardian(s). Exclusion Criteria
* GMFCS Level V (due to inability to cooperate with TMJ examination).
* History of craniofacial trauma, surgery, or congenital maxillofacial anomalies.
* Presence of neuromuscular diseases other than cerebral palsy.
* Active temporomandibular joint infection or acute systemic illness at the time of evaluation.
* Ongoing use of muscle relaxants or botulinum toxin injections in the jaw region within the past 6 months.
* Inability to complete the TMJ clinical examination due to behavioral or cognitive limitations.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of children and adolescents aged 6 to 18 years who have been clinically diagnosed with cerebral palsy (CP) and classified within Gross Motor Function Classification System (GMFCS) Levels I to IV. Participants will be recruited from pediatric neurology and physical therapy outpatient clinics of tertiary hospitals. The population is expected to represent a diverse range of CP subtypes (spastic, dyskinetic/ataxic, and mixed) and levels of functional motor impairment, allowing for subgroup analysis in relation to temporomandibular joint (TMJ) function. Participants must be able to comply with basic oral-motor assessments and have obtained informed consent from their parent(s) or legal guardian(s).
Sampling Method: Non-Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Temporomandibular Joint (TMJ) Functional Status | Single assessment at baseline
  Evaluation of TMJ functions using maximum mouth opening (mm), lateral jaw movement (mm), presence of joint sounds (click/crepitus), palpation tenderness, and Visual Analog Scale (VAS) for pain.

SECONDARY OUTCOMES:
Bruxism Prevalence | Single assessment at baseline
  Presence of bruxism identified through parental reports and clinical signs such as tooth wear and nocturnal grinding.
Gross Motor Function Level (GMFCS) | Single assessment at baseline
  Classification of motor function using GMFCS Levels I to IV to explore associations with TMJ dysfunction.
CP Subtype Distribution | Single assessment at baseline
  Classification of CP subtype as spastic, dyskinetic/ataxic, or mixed type to examine subgroup differences in TMJ outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri University, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No